CLINICAL TRIAL: NCT04618796
Title: Effect of COVID-19 Pandemic on Vaccination Compliance Among Children Attending Assiut University Children Hospital
Brief Title: Effect of COVID-19 Pandemic on Vaccination Compliance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Gamal Ahmed, Ressident doctor., Assiut University
Other Study IDs: Effect of COVID on vaccination
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Vaccine Refusal
Keywords: Covid19
MeSH Terms: conditions — Vaccination Refusal; COVID-19 | interventions — Vaccines

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: vaccine — Effect of COVID-19 pandemic on vaccination compliance among children attending Assiut University Children Hospital and what is the degree of that.

SUMMARY:
1- Evaluate the impact of the COVID-19 pandemic on pediatric vaccinations compliance among children attending to Assiut University Children Hospital ,assess the general health profile of studied children.

DETAILED DESCRIPTION:
Corona virus disease (COVID-19) is a disease caused by a new corona virus called Severe Acute Respiratory Syndrome Corona virus 2 (SARS-CoV-2). On March 11, the WHO Director-General declared COVID-19 a pandemic1. The first outbreak occurred in Wuhan, China. 2,3 COVID-19 pandemic has severely affected global health services.4 It is important not to overlook the value of some public health preventive interventions which cannot be postponed, such as vaccinations.5 As reported by WHO, the disruption of immunization services, even for brief periods, will result in increased numbers of susceptible individuals, raising the risks of an upsurge in outbreak-prone VPDs.6 The reduction of vaccination coverage could cause an increase in morbidity and mortality among children. Consequently, a greater burden could be placed on health systems. Examples from previous large epidemics (e.g. diphtheria in the former Soviet Union in 1990-1996 and in Venezuela in 2017-2018) show that, when vaccination coverage falls or vaccinations are disrupted, cases of infectious diseases that have disappeared can quickly re-emerge.7-8 Egypt declared a national state of emergency to control COVID-19 pandemic and implemented a stay-at-home order. Such strategies might result in decreased accessibility to routine immunization services, leaving children at risk for vaccine-preventable diseases and their complications.9 Great efforts are needed for rapid catch-up of children not up-to-date with routine vaccines. Parental concerns about potentially exposing their children to COVID-19 during vaccination visits might contribute to incompalince.10 Reminding parents of the vital need to protect their children against serious vaccine-preventable diseases is critical.

ELIGIBILITY:
Inclusion Criteria:

* Children from 12 to 24 months who admitted in Assiut University Children Hospital or attending the outpatient clinics

Exclusion Criteria:

* : Immunodeficiency (e.g chemotherapy, long term immunosuppressive therapy, hematologic tumor).

Ages: 1 Year to 2 Years | Sex: All
Age Groups: Child
Study Population: Children from 12 to 24 months
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Measure the vaccination coverage rate among the studied children after the COVID-19 pandemic | Baseline
  The investigators evaluate factors effect on compliance as covid-19, scioeconomic status, poverty, chronic disease and residance.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail lotfy, associated professor, Study Director — Assiut University; Mohamed Hamdy, professor, Study Director — Assiut University

REFERENCES:
- See also: Effect of COVID-19 pandemic on vaccination compliance among children attending Assiut University Children Hospital — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7419118/?fbclid=IwAR2wstjKh_FR2HQtHc1MSusCj_vlfpmNquWZJVEEbS1SXDX0KXR0gRTB4g4